CLINICAL TRIAL: NCT04194411
Title: Association of Plasma Biomarkers for Neurological Injury and Postoperative Delirium After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0925
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Delirium
Keywords: Neurofilament light; Tau; Delirium; Valvular heart surgery
MeSH Terms: conditions — Emergence Delirium; Charcot-Marie-Tooth disease, Type 1F; Pick Disease of the Brain; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for Nfl/Tau measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Valve surgery: Patients older than 65 years and undergoing elective valvular heart surgery

SUMMARY:
Delirium is one of the most common complications after cardiac surgeries, incidence of which is 20~70%. Causes and pathophysiology of delirium has not been elucidated yet, however, inflammatory response of the nervous system, imbalance of neurotransmitters and ischemia-reperfusion injury of brain tissue are thought to play a big role.

'Neurofilament light (Nfl)' and 'Tau' are proteins that comprise neurons, which are released into blood during acute brain injury. Increased serum concentrations of these markers are acknowledged to be associated with worse clinical outcomes in patients with acute brain injury. These proteins are also closely linked to degenerative changes in the nervous system and cognitive decline in Alzheimer's disease. Therefore, the increase in blood levels of 'Nfl' and 'Tau' may be related to the development of delirium.

The aim of this study is to investigate the association between 'Nfl' and 'Tau', serum markers of damage of the nervous system, and the development of delirium after cardiac surgery.

DETAILED DESCRIPTION:
1. Assessment of cognitive function and delirium Before the day before surgery, K-MMSE (Korean version of Mini-Mental State Exam) is conducted to check the subjects' baseline cognitive function.

   From the postoperative day 0 to 7, CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) for mechanically ventilated patients, or 3D-CAM (3-minute diagnostic assessment for delirium using the Confusion Assessment Method) for extubated patients is performed twice a day to assess whether delirium occurs. Records of the nurses are also checked.
2. Measurement of the serum levels of Nfl and Tau Serum concentrations of Nfl and Tau are measured after anesthetic induction, and at postoperative 6 hours

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing valvular heart surgery (>65 years old)

Exclusion Criteria:

* 1. Emergency operation
* 2. Patients with drug or alcohol abuse
* 3. Patients with major depressive disorder, major neurocognitive disorder or schizophrenia
* 4. Patients with schizophrenia
* 5. Patients who are not able to communicate verbally

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing valvular heart surgery (>65 years old)
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | Postoperative 7 days
  From the postoperative day 0 to 7, CAM-ICU (for mechanically ventilated patients) or 3D-CAM (for extubated patients) is performed twice a day. Electronic medical records of the patients are also assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea